CLINICAL TRIAL: NCT04803344
Title: The Effectiveness of Expressive Writing Intervention on the Psychological Wellness of the Mothers One Month After the Childbirth
Brief Title: The Effectiveness of Expressive Writing on a Sample of New Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Carlo Lai, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: URomLS_2
Record Dates: First submitted 2020-11-26; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Maternal Distress; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): After the childbirth, writing group participants has been asked to write for 3 consecutive days, 20 minutes each days, all the deepest emotions and feelings related to the pregnancy.
  Interventions: Behavioral: Expressive Writing tecnique
- Control Group (Active Comparator)
  Interventions: Behavioral: Neutral Writing

INTERVENTIONS:
Behavioral: Expressive Writing tecnique — Expressive Writing (EW), is a simple, potentially inexpensive, therapeutic intervention which involves writing daily for 15-20 min over 3-4 consecutive days. EW can be completed at home without the need for facilitation, a specialist therapist or a dedicated facility.
  Arms: Experimental Group
Behavioral: Neutral Writing — Participants were asked to write on neutral objects or events.
  Arms: Control Group

SUMMARY:
This pilot study aims to evaluate the effects of an expressive writing intervention on a sample of new mothers after the childbirth on the psychological health and on the healthcare costs. The mothers were evaluated also in a follow-up one month after the end of the expressive writing intervention.

DETAILED DESCRIPTION:
Women are recruited starting from the sixth month of pregnancy; forty-one eventually agreed to participate and they were randomly assigned to two groups: an Experimental group (treated with the expressive writing task, one weeks-three months after childbirth) and a Control group (no intervention).

Psychological health is measured at three stages:

before intervention, at 8-9 months pregnant (T0); after intervention, from 1 week to 3 months after delivery (T1); and a follow-up after 1 to 3 months (T2). The assessment protocol consists of the Attachment Style Questionnaire (ASQ), the Prenatal Attachment Inventory (PAI), the Toronto Alexythimia Scale-20 (TAS-20), the Beck Depression Inventory (BDI-13), the State-Trait Anxiety Inventory (STAI-Y), the Rating Scale For Rapid Stress Assessment (VRS) and the 12-Item Short Form Survey (SF-12). The healthcare costs are collected at baseline (T0) and follow-up (T2) with a survey created ad hoc, in which participants reported the number and the type of the medical examinations, hospitalisations, prescribed drugs etc. Social and personal data are collected from the first survey.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* > 6 months of pregnancy
* no medical complications during pregnancy

Exclusion Criteria:

* medical complication during pregnancy
* no comprehension of Italian language

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study was conducted on new mothers
Enrollment: 41 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Before (T0) and after the writing intervention (T1) and at the follow-up (T2). The outcome assessment lasts about 1 hour
  In order to evaluate the Health-related quality of life, the 12-Item Short Form Health Survey was used. This standardized questionnaire is composed by 12 items selected from SF-36 and produces two summaries, physical (PCS) and mental (MCS) scale (Brazier and Roberts, 2004).
Anxiety | Before (T0) and after the writing intervention (T1) and at the follow-up (T2). The outcome assessment lasts about 1 hour
  In order to evaluate the levels of anxiety, the Spielberger State-Trait Anxiety Inventory, STAI-Y, (Spielberger, 1983; Spielberger et al., 1970) was used. It is a self-report questionnaire developed to evaluate both state and trait anxiety, respectively a transitory emotional state and a personality trait considered relatively stable.
Depression | Before (T0) and after the writing intervention (T1) and at the follow-up (T2). The outcome assessment lasts about 1 hour
  In order to evaluate the levels of depression, The 13-item short form of Beck Depression Inventory (BDI-II) was used.
Healthcare spending | Before (T0) and after the writing intervention (T1) and at the follow-up (T2). The outcome assessment lasts about 1 hour
  In order to test the healthcare spending to all participants were asked (through a specific questionnaire built ad hoc for the specific situation) the number of medical visits, the number of hospitalizations, the number of admissions to emergency room for acute episodes, the number of hospitalizations stay days in the last year. The study hypothesized a lower number of medical visits, hospitalization's days and admissions to emergency room for those mothers who performed the expressive writing task.
Stress | Before (T0) and after the writing intervention (T1) and at the follow-up (T2). The outcome assessment lasts about 1 hour
  In order to test the stress levels, the Valutazione Rapida dello stress (VRS) was used. The VRS is rapid self-assessment rating scale for measure of percieved stress. This scale is composed of 15 items and five areas: anxiety, depression, somatization, aggressiveness, and social support. The social support scale measures the percieved lack of social support (Tarsitani and Biondi, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lai, Professor, Principal Investigator — Sapienza university of Rome, Department of Dynamic and Clinical Psychology, and Health Studies
Locations (1):
- Department of Dynamic and Clinical Psychology, and Health Studies, Sapienza University, Rome, Italy

IPD SHARING:
Plan to Share IPD: No